CLINICAL TRIAL: NCT01116323
Title: Emergency Department Crowding in Relation to In-hospital Adverse Medical Events
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Verelst Sandra, MD, KU Leuven
Other Study IDs: AE1.7.005.11.N.00
Record Dates: First submitted 2010-05-03; First posted 2010-05-04 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Adverse Effects
Keywords: Adverse events; Adverse effects; Emergency Service, Hospital; Emergency department; Crowding
MeSH Terms: conditions — Emergencies; Crowding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — None Retained - no samples retained
Oversight: Data Monitoring Committee: No

SUMMARY:
Since the report "To Err is Human" by the Institute of Medicine (IOM) in 1999, attention was brought to the general public that adverse events in medicine are common and are one of the leading causes of morbidity and mortality within the United States. The report estimates that 44,000 - 98,000 patients hospitalized in the United States die each year as a result of medical errors.

In spite of the growing patient safety movement worldwide, health care has not become measurably safer. Health care is one of the few risk-prone areas in which public demand limits the use of common-sense safety-enhancing solutions, such as limiting the flow and choosing the type of incoming patients. The latter is especially true for emergency departments (EDs) since they deliver an important public service by providing emergency care 24 hours a day, 365 days per year, without discrimination by social or economic status. One of the key expectations of EDs is the ability to provide immediate access and stabilization for those patients who have an emergency medical condition. However, emergency department (ED) crowding is recognized to be a major, international problem that affects patients and providers. A recent report from the IOM noted that the increasing strain caused by crowding is creating a deficit in quality of emergency care. Crowding has been associated with reduced access to emergency medical services, delays in care for cardiac patients, increased patient mortality, inadequate pain management, increased costs of patient care, and delays in administration of antibiotic therapy.

Several issues remain concerning ED crowding and it's relation to adverse events. First, the existing evidence on adverse event occurrence during ED crowding is largely anecdotal and inconclusive. Secondly, although a few studies showed a relationship between ED crowding and mortality, neither of these examined the causes of excess mortality. Finally, although a significant increase in the average length of hospital stay was shown during ED crowding the reasons for this are open to speculation.

The purpose of this study therefore is to identify six explicit adverse events and mortality for patients who were admitted through ED and to compare these results in relation to ED crowding. This will provide us novel insight into the reasons for the hypothesized increased mortality during ED crowding.

DETAILED DESCRIPTION:
Since "ED crowding" is an unplanned condition, a randomized controlled trial is not possible to assess its impact on adverse patients' outcome. Therefore, a large prospective cohort study, with careful matching and correcting for risk factors is the second best design.

The ED occupancy rate, defined as the ratio of the total number of ED patients to the number of licensed treatment bays per hour, will be used as a measure of ED crowding. The numerator includes all patients in the ED at any point during each study hour, regardless of ED location (including in the waiting room, boarding, hallway location). The denominator, constant per study hour, includes the total number of licensed treatment bays as defined according to the ED's original blueprint but excludes hallway locations. For each hour of the day, the ED occupancy rate will be derived from the ED information system. 104 weeks are divided into 13-week seasonal blocks and nursing shifts starting 23:00, 07:00 and 15:00. The mean ED occupancy rate is calculated for each shift as the sum of the occupancy rates within that shift divided by 8. The top quartile of all mean ED occupancy rates during the cohort period is considered as crowded. In order to match both 'crowded 'and 'not crowded' cohorts, the following data elements are extracted from the hospital information system for each registered patient: demographic data (age, sex, co-morbidities); referral source, surgical or medical admission; time of arrival (including season, month of year, day of week, time of day); triage category; ED and total hospital length of stay; and final admission diagnosis.

Medical records of patients who presented to the ED will be reviewed for the occurrence of six adverse events and mortality up to ten days of their ED stay. The six adverse events are searched through explicit clinical criteria. The reviewer first rates on a scale of 1 to 6 the confidence that medical management caused an adverse event. If the rating is 5 or 6, indicating that the injury is probably or definitely caused by management, the event is considered an adverse event. The same rating score is used to assess the degree of preventability. Hospital mortality will be searched for all patients who presented to the ED at some point in time and died during that hospital stay.

In order to identify an adverse event occurrence hazard ratio of 1.2 with a power of 0.9 during ED crowding, a cohort of 104,000 patients is needed. Therefore, data will be retrieved during a 2 year period during which the reviewer is blinded to the degree of ED crowding in relation to the findings on adverse events. The occurrence of adverse events and mortality will be compared to not crowded shifts, corrected for baseline risk factors. A carefully standardized admission form for registration of relevant information as well as a computerized search tool for screening for adverse events will allow finalizing this study within the foreseen time frame.

ELIGIBILITY:
Inclusion Criteria:

* All adult (18 years or older) patients presenting to the ED
* All adult (18 years or older) patients transferred from the ward to ED for upgrading of care

Exclusion Criteria:

* All patients who died on arrival in the ED
* Patients transferred from another acute care facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (18 years or older) patients presenting to the ED
Sampling Method: Probability Sample
Enrollment: 104000 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of six adverse events | During the 2 year period of prospective study, the occurrence of 6 adverse events will be searched from the time to ED admission up to 10 days after discharge from ED
  Search for either hospital acquired pneumonia, deep venous thrombosis/pulmonary embolism, sepsis, acute renal failure, shock/cardiac arrest, or gastrointestinal hemorrhage/gastric ulcer through explicit clinical criteria.

SECONDARY OUTCOMES:
Mortality | During the 2 year period of prospective study, mortality will be searched from the time to ED admission until hospital discharge of the patient
  Hospital mortality
ED length of stay | Whole ED stay
  Time from ED admission until discharge home or to hospital ward
Hospital length of stay | Whole hospital stay
  Time from hospital admission until hospital discharge
Time to antibiotics administration in case of pneumonia | Whole ED stay
  Time (in hours and minutes) to administration of antibiotics in case a diagnosis of pneumonia is made in the ED

CONTACTS AND LOCATIONS:
Overall Officials: Greet Van den Berghe, MD, Ph D, Principal Investigator — Catholic University Leuven
Locations (1):
- Emergency Department, Catholic University Leuven, Leuven, Vlaams Brabant, Belgium

REFERENCES:
- [Background] Richardson DB. Increase in patient mortality at 10 days associated with emergency department overcrowding. Med J Aust. 2006 Mar 6;184(5):213-6. doi: 10.5694/j.1326-5377.2006.tb00204.x. PMID 16515430